CLINICAL TRIAL: NCT02964910
Title: An Open, Pared Trial of Recombinant Hepatitis E Vaccine (Escherichia Coli) Hecolin® in the Chronic Hepatitis B Patients on the Clinical Stability .( Aged 30 Years or Over)
Brief Title: A Phase Ⅳ Clinical Trial of the Recombinant Hepatitis E Vaccine (Escherichia Coli)(the Chronic Hepatitis B Patients )
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiamen Innovax Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-HE-009
Record Dates: First submitted 2016-11-09; First posted 2016-11-16 (Estimated); Results first posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis E
Keywords: Hepatitis E
MeSH Terms: conditions — Hepatitis E | interventions — hecolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the chronic Hepatitis B patients (Experimental): Participants in this arm are aged over 30 years and would receive three doses of Recombinant Hepatitis E Vaccine (Escherichia Coli)(Hecolin®) at 0,1,6 month.
  Interventions: Biological: Recombinant Hepatitis E Vaccine (Escherichia Coli)
- the healthy volunteer (Active Comparator): Participants in this arm are aged over 30 years and would receive three doses of Recombinant Hepatitis E Vaccine (Escherichia Coli)(Hecolin®) at 0,1,6 month.
  Interventions: Biological: Recombinant Hepatitis E Vaccine (Escherichia Coli)

INTERVENTIONS:
Biological: Recombinant Hepatitis E Vaccine (Escherichia Coli) — Participants would receive 3 doses of Recombinant Hepatitis E Vaccine (Escherichia Coli) intramuscularly at 0, 1, 6 month.
  Other Names: Hecolin®

SUMMARY:
This phase IV clinical study was designed to evaluate the immunogenicity and safety of Hecolin® in the chronic Hepatitis B patients on the clinical stability.

DETAILED DESCRIPTION:
This phase IV clinical study was designed to evaluate the immunogenicity and safety of the recombinant Hepatitis E vaccine(Hecolin®), manufactured by Xiamen Innovax Biotech CO., LTD., in the chronic Hepatitis B patients on the clinical stability and aged over 30 years of age at enrollment. The study volunteers will receive the 3 doses of Hecolin® administered intramuscularly according to a 0-1-6 month schedule.

ELIGIBILITY:
Inclusion Criteria(all volunteers):

1. Aged over 30 years old on the day of enrollment
2. Axillary temperature is below than 37.0 ℃.
3. No administration of HEV vaccine before the study
4. Judged as healthy and eligible for vaccination by the investigators through a selfreported medical history and some physical examinations.
5. Able to understand this study information and willing to comply with all study requirements.
6. Willing to participate in this study and sign informed consent form.
7. Negative serological markers for hepatitis E

Inclusion Criteria(experiment group):

1. ALT < 1.5×ULN
2. No spleen swelling,no cirrhosis and no hepatocellular carcinoma

Inclusion Criteria(control group):

1. HBsAg(-)

Exclusion Criteria:

1. With clinical evidence of malignant tumor
2. History of severe cardio-cerebrovascular disease
3. Administration of hepatotoxicity drugs before or during the study
4. Pregnancy,breast-feeding or plan to be pregnant in 7 months later
5. Participated in any other clinical trial during the study period.
6. Use of any investigational product or non-registered product (drug or vaccine)within 30 days preceding the first dose of the study vaccine or plan to use during the study period.
7. Received immunosuppressed, immunoregulation therapy or corticosteroid systemic therapy for more than 14 days in the 6 months before entry, except local treatment.
8. Administration of any immunoglobulin or blood products within 3 months preceding the first dose of the study vaccine,or plan to use during the study period.
9. Administration of any inactivated vaccines within 14 days preceding the first dose of the study or attenuated live vaccines within 21 days preceding the first dose of the study.
10. Had a fever (axillary temperature over 38°C) within 3 days or acute illness requiring systemic antibiotics or antiviral treatment within 5 days before vaccination.
11. Immunodeficiency (such as HIV carriers), primary disease of important organs, malignant tumor, or any immune disease (such as systemic lupus erythematosus, arthritis pauperum, splenectomy or functional asplenia or other disease which might affect immune response).
12. History of allergic disease or history of serious adverse events occurring after vaccination, i.e., allergy,urticaria, dyspnea, angioneurotic edema or abdominal pain.
13. Allergic history to any component of this vaccine.
14. Asthma that needed emergency treatment, hospitalization, oral or intravenous corticosteroid to keep stable in the past two years.
15. Combining another severe internal medicine disease(such as severe hypertension, cardiopathy,diabetes and hyperthyroidism)
16. Anomal coagulation function or coagulopathy diagnosed by doctor
17. Epilepsy(not including alcohol epilepsy within 3 years prior to abstinence and simple epilepsy that do without curing within 3 years prior to the study )
18. Anomal psychology or mind affecting the individual's ability to obey the study requie
19. Other medical, psychological, social or occupational factors that, according to the investigators' judgment,might affect the individual's ability to obey the protocol or sign the informed consent.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aiqiang Xu, Principal Investigator — Shandong Provincial Center for Disease Control and Prevention
Locations (1):
- Rushan Center for Disease Control and Prevention, Weihai, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- the Chronic Hepatitis B Patients; the Healthy Volunteer: Participants in this arm are aged over 30 years and would receive three doses of Recombinant Hepatitis E Vaccine (Escherichia Coli)(Hecolin®) at o,1,6 month.
  Recombinant Hepatitis E Vaccine (Escherichia Coli): Participants would receive 3 doses of Recombinant Hepatitis E Vaccine (Escherichia Coli) intramuscularly at 0, 1, 6 month.
Period: Overall Study
Arm/Group | the Chronic Hepatitis B Patients | the Healthy Volunteer
Started | 235 | 240
Completed | 192 | 196
Not Completed | 43 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | the Chronic Hepatitis B Patients | the Healthy Volunteer | Total
Number analyzed (Participants) | 235 | 240 | 475
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (9.7) | 53.4 (9.5) | 53.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 97 | 193
  Male | 139 | 143 | 282
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whose Anti-HEV Antibody Seroconverted at One Month After The Third Dose
Description: Measure the number of participants whose anti-HEV antibody seroconverted at month 7 to evaluate the immunogenicity of the Hepatitis E vaccine.
Time Frame: Month 7
Population: Totally 192 CHB participants and 196 healthy participants were involved in per-protocol set, who meet the meet the requirements 1) whole-course inoculation, 2)having the results of anti-HEV antibody test before and after immunization, 3) anti-HEV antibody negative before immunization.
Measure: Count of Participants; unit: Participants
Arm/Group | the Chronic Hepatitis B Patients | the Healthy Volunteer
Number analyzed (Participants) | 192 | 196
Participants | 188 | 196
Statistical Analysis 1: Comparison: the Chronic Hepatitis B Patients vs the Healthy Volunteer; Test type: Non-Inferiority — The criteria of the immunogenicity non-inferiority between CHB group and healthy adults group were: the lower limit of 95% CI of the seroconversion rate difference was not less than -10%; the seroconversion rate difference(%) = -2.08, 95% CI 2-sided [-5.23 to 0.22]

2. Primary Outcome: Geometric Mean Concentrations of Anti-HEV Antibody at One Month After The Third Dose
Description: Measure the level of anti-HEV antibody in serum samples at month 7 to evaluate the immunogenicity of the Hepatitis E vaccine.
  Wu/ml：World Health Organization (WHO) units per ml. The WHO standard was used to calibrate the antibody quantitative reference.
Time Frame: Month 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Wu/ml
Arm/Group | the Chronic Hepatitis B Patients | the Healthy Volunteer
Number analyzed (Participants) | 192 | 196
Wu/ml | 11.89 [9.86 to 14.35] | 17.35 [15.57 to 19.34]
Statistical Analysis 1: Comparison: the Chronic Hepatitis B Patients vs the Healthy Volunteer; Test type: Non-Inferiority — The criteria of the immunogenicity non-inferiority between CHB group and healthy adults group were: the lower limit of 95%CI of the GMC ratio was not lower than 0.5; GMC ratio = 0.69, 95% CI 2-sided [0.55 to 0.85]

3. Secondary Outcome: Number of Participants With Changes in Liver Function Index Before and One Month After the First Dose
Description: ALT, AST and TBIL were detected in both groups to determine the liver function of participants. The grade of ALT, AST and TBIL was determined according to the rules issued by CFDA. The fluctuations were classified into three categories: "no change" indicated no grade change; "processed" indicated a change from normal to abnormal or an increase in grade; and "improved" indicated a change from abnormal to normal or a decrease in grade or the change from abnormal to normal.
Time Frame: Day 0-Month 1
Population: All the participants who visited at one month after the first dose.
Measure: Count of Participants; unit: Participants
Arm/Group | the Chronic Hepatitis B Patients | the Healthy Volunteer
Number analyzed (Participants) | 223 | 220
Participants
  ALT: no change | 208 | 215
  ALT: processed | 5 | 4
  ALT: improved | 10 | 1
  AST: no change | 186 | 211
  AST: processed | 18 | 5
  AST: improved | 19 | 4
  TBIL: no change | 184 | 169
  TBIL: processed | 12 | 25
  TBIL: improved | 27 | 26

4. Secondary Outcome: Number of Participants With Changes in Liver Function Index Before and One Month After the Third Dose
Description: as for outcome 3
Time Frame: Month 6-Month 7
Population: All the participants who visited at one month after the third dose.
Measure: Count of Participants; unit: Participants
Arm/Group | the Chronic Hepatitis B Patients | the Healthy Volunteer
Number analyzed (Participants) | 213 | 206
Participants
  ALT: no change | 204 | 206
  ALT: processed | 2 | 0
  ALT: improved | 7 | 0
  AST: no change | 178 | 203
  AST: processed | 8 | 2
  AST: improved | 27 | 1
  TBIL: no change | 182 | 195
  TBIL: processed | 6 | 1
  TBIL: improved | 25 | 10

5. Secondary Outcome: Number of Participants With Changes in Liver Function Index Before The First Dose and One Month After the Third Dose
Description: as for outcome 3
Time Frame: Day0-Month 7
Population: All the participants who visited at one month after the third dose.
Measure: Count of Participants; unit: Participants
Arm/Group | the Chronic Hepatitis B Patients | the Healthy Volunteer
Number analyzed (Participants) | 213 | 206
Participants
  ALT: no change | 199 | 204
  ALT: processed | 1 | 0
  ALT: improved | 13 | 2
  AST: no change | 177 | 200
  AST: processed | 8 | 2
  AST: improved | 28 | 4
  TBIL: no change | 175 | 162
  TBIL: processed | 5 | 1
  TBIL: improved | 33 | 43

6. Secondary Outcome: Number of Participants Who Experienced Any Adverse Reactions/Events
Description: Any adverse reactions/events contains solicited and unsolicited adverse reactions/events during the whole period of observation.
Time Frame: Day 0-Month 7
Population: All the participants who received at least one injection.
Measure: Count of Participants; unit: Participants
Arm/Group | the Chronic Hepatitis B Patients | the Healthy Volunteer
Number analyzed (Participants) | 235 | 240
Participants | 92 | 97
Statistical Analysis 1: Comparison: the Chronic Hepatitis B Patients vs the Healthy Volunteer; Test type: Other — The differences in incidence rate of ADR\AE between the two groups were compared; p = 0.778, Chi-squared

7. Secondary Outcome: Number of Participants Who Experienced Solicited Adverse Reactions/Events
Description: Number of participants who experienced local, system adverse reactions/events within 7 days after each vaccination.
Time Frame: Day 0-Day 7
Population: All the participants who received at least one injection.
Measure: Count of Participants; unit: Participants
Arm/Group | the Chronic Hepatitis B Patients | the Healthy Volunteer
Number analyzed (Participants) | 235 | 240
Participants | 42 | 40
Statistical Analysis 1: Comparison: the Chronic Hepatitis B Patients vs the Healthy Volunteer; Test type: Other — The differences in incidence rate of ADR\AE between the two groups were compared; p = 0.728, Chi-squared

8. Secondary Outcome: Number of Participants Who Experienced Solicited Local Adverse Reactions/Events
Description: Number of participants who experienced solicited local adverse reactions/events within 7 days after each vaccination.
Time Frame: Day 0-Day 7
Population: All the participants who received at least one injection.
Measure: Count of Participants; unit: Participants
Arm/Group | the Chronic Hepatitis B Patients | the Healthy Volunteer
Number analyzed (Participants) | 235 | 240
Participants | 17 | 17
Statistical Analysis 1: Comparison: the Chronic Hepatitis B Patients vs the Healthy Volunteer; Test type: Other — The differences in incidence rate of ADR\AE between the two groups were compared; p = 0.949, Chi-squared

9. Secondary Outcome: Number of Participants Who Experienced Solicited System Adverse Reactions/Events
Description: Number of participants who experienced solicited system adverse reactions/events within 7 days after each vaccination.
Time Frame: Day 0-Day 7
Population: All the participants who received at least one injection.
Measure: Count of Participants; unit: Participants
Arm/Group | the Chronic Hepatitis B Patients | the Healthy Volunteer
Number analyzed (Participants) | 235 | 240
Participants | 31 | 28
Statistical Analysis 1: Comparison: the Chronic Hepatitis B Patients vs the Healthy Volunteer; Test type: Other — The differences in incidence rate of ADR\AE between the two groups were compared; p = 0.614, Chi-squared

10. Secondary Outcome: Number of Participants Who Experienced Unsolicited Adverse Reactions/Events
Description: Number of participants who experienced unsolicited adverse reactions/events during the whole period of observation.
Time Frame: Day 0-Month 7
Population: All the participants who received at least one injection.
Measure: Count of Participants; unit: Participants
Arm/Group | the Chronic Hepatitis B Patients | the Healthy Volunteer
Number analyzed (Participants) | 235 | 240
Participants | 68 | 70
Statistical Analysis 1: Comparison: the Chronic Hepatitis B Patients vs the Healthy Volunteer; Test type: Other — The differences in incidence rate of ADR\AE between the two groups were compared; p = 0.956, Chi-squared

ADVERSE EVENTS:
Time Frame: 0-7 months
Description: The definitions of "All-Cause Mortality","Serious Adverse Events" and "Adverse Events" are consistent with the clinicaltrials.gov Definitions.
  One death was due to myocardial infarction.
Arm/Group | the Chronic Hepatitis B Patients | the Healthy Volunteer
All-Cause Mortality (participants affected / at risk) | 1/235 | 0/240
Serious Adverse Events (participants affected / at risk) | 6/235 | 2/240
Other Adverse Events (participants affected / at risk) | 15/235 | 19/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | the Chronic Hepatitis B Patients (N=235) | the Healthy Volunteer (N=240)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) — Grade 3: SBP≥180mmHg and\or DBP≥110mmHg
subacute thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
VertebrobasilarArtery Insufficiency (Nervous system disorders) | 1 (1) | 1 (1)
lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | the Chronic Hepatitis B Patients (N=235) | the Healthy Volunteer (N=240)
pyrexia (General disorders) | 15 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT02964910/Prot_SAP_000.pdf